CLINICAL TRIAL: NCT05366881
Title: cfDNA Assay Multicenter Prospective Observational Validation for Early Cancer Detection, Minimal Residual Disease, and Relapse
Brief Title: cfDNA Assay Prospective Observational Validation for Early Cancer Detection and Minimal Residual Disease
Acronym: CAMPERR
Status: Recruiting | Type: Observational
Sponsor: Adela, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: Adela-EDMRD-001
Record Dates: First submitted 2022-05-03; First posted 2022-05-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Brain Cancer; Breast Cancer; Bladder Cancer; Cervical Cancer; Colorectal Cancer; Endometrial Cancer; Esophageal Cancer; Stomach Cancer; Head and Neck Cancer; Hepatobiliary Cancer; Leukemia; Lung Cancer; Lymphoma; Multiple Myeloma; Ovarian Cancer; Pancreatic Cancer; Prostate Cancer; Renal Cancer; Sarcoma; Thyroid Cancer
Keywords: Multi-cancer early detection; Liquid Biopsy; Methylome; Cancer screening; cell-free DNA
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Leukemia; Lung Neoplasms; Lymphoma; Multiple Myeloma; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Kidney Neoplasms; Sarcoma; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and extracted cell-free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cases will include participants with newly diagnosed, treatment-naive cancer at the time of enrollment.
- Controls: Controls will include participants without known cancer at the time of enrollment.

SUMMARY:
This is an observational case-control study to train and validate a genome-wide methylome enrichment platform to detect multiple cancer types and to differentiate amongst cancer types. The cancers included in this study are brain, breast, bladder, cervical, colorectal, endometrial, esophageal, gastric, head and neck, hepatobiliary, leukemia, lung, lymphoma, multiple myeloma, ovarian, pancreatic, prostate, renal, sarcoma, and thyroid. These cancers were selected based on their prevalence and mortality to maximize impact on clinical care.

Additionally, the ability of the whole-genome methylome enrichment platform to detect minimal residual disease after completion of cancer treatment and to detect relapse prior to clinical presentation will be evaluated in lung cancer. This cancer was selected based on the existing clinical landscape and treatment availability.

DETAILED DESCRIPTION:
This is an observational case-control study that includes individuals with cancer and individuals without known cancer. All participants will have clinical follow-up after enrollment. A subset of individuals with cancer will also have longitudinal blood sampling to evaluate the ability of the genome-wide methylome enrichment platform to detect minimal residual disease. This includes individuals with Stage I-III lung cancer (Tier 1 Cancers).

At baseline, all participants will provide a blood sample and applicable clinical data.

Participants with a Tier 1 cancer will have clinical follow-up and blood draws after the completion of first-line treatment, every 3 months for the first year after first-line treatment, and every 6 months for an additional 2 years. All other cases may have clinical follow-up once a year for 3 years after enrollment.

Control participants will have clinical follow-up every 6 months for up to 3 years from enrollment to evaluate cancer status.

The blood test to be used in this study is a highly sensitive, epigenomic-based genome-wide methylome enrichment platform. The assay includes bisulfite-free, non-degradative genome-wide DNA methylation profiling from small quantities of cell-free DNA (cfDNA). Libraries constructed from cfDNA are enriched for methylated CpGs and preserve the native fragment length. This is followed by high throughput sequencing.

For all assays, samples from participants with cancer and participants without cancer will be run together to reduce batch effects using methodology determined by the Sponsor. Results from the liquid biopsy test will not be returned to clinicians or participants.

ELIGIBILITY:
Case Inclusion Criteria:

* Newly diagnosed (within 120 days) with cancer or a recurrence of a cancer diagnosed >5 years ago of one of the following subtypes: Invasive Brain, Breast, Bladder, Cervical, Colorectal, Endometrial, Esophageal, Gastric, Head and Neck, Hepatobiliary, Lung, Ovarian, Pancreatic, Prostate, Renal, Sarcoma, Thyroid; Leukemia, Lymphoma, Multiple Myeloma
* Able and willing to provide informed consent
* ≥40 years of age

Case Exclusion Criteria:

* Currently receiving any treatment for cancer
* Currently taking any demethylating agents/DNA hypomethylating agents
* Simultaneously diagnosed with two or more invasive cancers
* Diagnosed with any invasive or non-invasive cancer in addition to the index cancer in the last 5 years
* Currently diagnosed with any chronic hematopoietic cancer (e.g. chronic CLL) in addition to the index cancer
* Currently diagnosed with any myelodysplastic syndromes and/or precursor hematologic conditions (e.g. MGUS) in addition to the index cancer
* Women who are known to be pregnant (self-reported)

Control Inclusion Criteria

* Not diagnosed with any cancer in the last 5 years (non-invasive cancer is allowed)
* Able and willing to provide informed consent
* ≥40 years of age

Control Exclusion Criteria

* Currently receiving any treatment for cancer
* Currently taking any demethylating agents/DNA hypomethylating agents
* Women who are known to be pregnant (self-reported)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll individuals with newly diagnosed cancer as cancer cases and individuals without known cancer as controls. Participants will be enrolled from sites across the United States.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Detection of cancer | 24 months
  Differentiation of cancer signals from cases and non-cancer signals from controls based on analysis of cfDNA using the genome-wide methylome enrichment platform

SECONDARY OUTCOMES:
Detection of specific cancer types | 24 months
  Differentiation of cancer signals from cases with a specific cancer type and non-cancer signals from controls based on analysis of cfDNA using the genome-wide methylome enrichment platform
Tissue of origin | 18 months
  Identification of the correct tissue of origin (as determined by clinical diagnosis) for cancer cases based on analysis of cfDNA using the genome-wide methylome enrichment platform
Clinical outcomes | 54 months
  Recurrence-free survival and overall survival among cancer cases

CONTACTS AND LOCATIONS:
Overall Officials: Brian Rini, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (17):
- United States (17):
  - City of Hope, Duarte, California
  - Miami Cancer Institute, Miami, Florida
  - North Georgia Health System, Gainesville, Georgia
  - Baptist Floyd, New Albany, Indiana
  - Baptist Corbin, Corbin, Kentucky
  - Baptist Hardin, Elizabethtown, Kentucky
  - Baptist Lexington, Lexington, Kentucky
  - Baptist Paducah, Paducah, Kentucky
  - Allina Health Cancer Institute, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - McLeod Health, Florence, South Carolina
  - Baptist (BHMCC), Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Elligo Health Research, Inc., Austin, Texas